CLINICAL TRIAL: NCT02348762
Title: Energetics and Function in Older Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Rajagopal V Sekhar, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-34686 Glutathione and Aging
Record Dates: First submitted 2015-01-15; First posted 2015-01-28 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Aging; Erythrocyte Glutathione Deficiency; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness | interventions — Cysteine; Glycine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glycine and N-acetylcysteine (Experimental): Older subjects will be studied before and after taking oral cysteine (as n-acetylcysteine) and glycine for 6 months
  Interventions: Dietary Supplement: Cysteine (as n-acetylcysteine) and Glycine

INTERVENTIONS:
Dietary Supplement: Cysteine (as n-acetylcysteine) and Glycine — Older subjects will be studied before and after receiving cysteine and glycine

SUMMARY:
The investigators have previously reported that older patients with HIV are deficient in glutathione (GSH) due to decreased availability of cysteine and glycine, and that oral supplementation with cysteine (as n-acetylcysteine) and glycine for 2-weeks corrects their own levels, and improves concentrations of red-cell GSH. The investigators also found that when GSH deficient, subjects had impaired mitochondrial energetics and this improved with an increase in intracellular GSH concentrations. The current proposal will investigate if cysteine and glycine supplementation for a duration of 24 weeks will result in changes in : (a) GSH levels; (b) body composition/anthropometry; (c) strength and function; (d) quality of life; (e) mitochondrial energetics; (f) biochemistry (including dyslipidemia and oxidative stress); (g) protein and glucose metabolism; (h) cognition and memory. 3 months after completing supplementation, measurement of GSH concentrations, strength, function, mitochondrial energetics and neurocognitive tests will be done to determine the effects of washout.

DETAILED DESCRIPTION:
Data not available at present

ELIGIBILITY:
Inclusion Criteria:

Older subjects:

* age 70-80 years;

Younger subjects:

* age 21-30 years

Exclusion Criteria:

1. No known diabetes, liver disease, kidney disease, coronary heart disease, stroke, or cancer;
2. Any limitations in ability to walk;
3. Triglyceride concentrations greater than 500 mg/dl (if lipid lowering medications are stopped);
4. BMI less than 20.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11; Primary Completion 2018-11 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Red blood cell concentrations of Glutathione measured by HPLC | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: R V Sekhar, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor Metabolic Research Unit (MRU), Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No